CLINICAL TRIAL: NCT03674710
Title: A Multi-center, Prospective, Single-blind, Controlled Trial Comparing Suction Technique, Slow-pull Method and Wet Suction Technique on Specimen Quality and Diagnostic Accuracy in Endoscopic Ultrasound-guided Fine-needle Aspiration
Brief Title: A Multi-center, Prospective, Single-blind, Controlled Trial Comparing Diagnostic Value of Different EUS-FNA Techniques
Acronym: EUS-FNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: B2017-195
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Neoplasms; Infection; Inflammation; Lymphoma; Cancer; Sarcoid; Mass Lesion
Keywords: EUS-FNA
MeSH Terms: conditions — Neoplasms; Infections; Inflammation; Lymphoma; Sarcoidosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A (Experimental): Patients assigned to group A will be sampled for a total of 3 consecutive FNA passes with a sequential method of "standard suction", "slow-pull", and "wet suction". After completing all the passes, the obtained specimen will be packed individually and sent to pathologists who are blind to the method sequence.
  Interventions: Procedure: Standard suction, slow-pull, wet suction
- Group B (Experimental): Patients assigned to group B will be sampled for a total of 3 consecutive FNA passes with a sequential method of "standard suction", "wet suction", and "slow-pull". After completing all the passes, the obtained specimen will be packed individually and sent to pathologists who are blind to the method sequence.
  Interventions: Procedure: Standard suction, wet suction, slow-pull
- Group C (Experimental): Patients assigned to group C will be sampled for a total of 3 consecutive FNA passes with a sequential method of "slow-pull", "standard suction", and "wet suction". After completing all the passes, the obtained specimen will be packed individually and sent to pathologists who are blind to the method sequence.
  Interventions: Procedure: Slow-pull, standard suction, wet suction
- Group D (Experimental): Patients assigned to group D will be sampled for a total of 3 consecutive FNA passes with a sequential method of "slow-pull", "wet suction", and "standard suction". After completing all the passes, the obtained specimen will be packed individually and sent to pathologists who are blind to the method sequence.
  Interventions: Procedure: Slow-pull, wet suction, standard suction
- Group E (Experimental): Patients assigned to group E will be sampled for a total of 3 consecutive FNA passes with a sequential method of "wet suction", "standard suction", and "slow-pull". After completing all the passes, the obtained specimen will be packed individually and sent to pathologists who are blind to the method sequence.
  Interventions: Procedure: Wet suction, standard suction, slow-pull
- Group F (Experimental): Patients assigned to group F will be sampled for a total of 3 consecutive FNA passes with a sequential method of "wet suction", "slow-pull", and "standard suction". After completing all the passes, the obtained specimen will be packed individually and sent to pathologists who are blind to the method sequence.
  Interventions: Procedure: Wet suction, slow-pull, standard suction

INTERVENTIONS:
Procedure: Standard suction, slow-pull, wet suction — Patients will be sampled for a total of 3 consecutive FNA passes with a sequential method of "standard suction", "slow-pull", and "wet suction". After completing all the passes, the obtained specimen will be packed individually and sent to pathologists who are blind to the method sequence.
  Arms: Group A
Procedure: Standard suction, wet suction, slow-pull — Patients will be sampled for a total of 3 consecutive FNA passes with a sequential method of "standard suction", "wet suction", and "slow-pull". After completing all the passes, the obtained specimen will be packed individually and sent to pathologists who are blind to the method sequence.
  Arms: Group B
Procedure: Slow-pull, standard suction, wet suction — Patients will be sampled for a total of 3 consecutive FNA passes with a sequential method of "slow-pull", "standard suction", and "wet suction". After completing all the passes, the obtained specimen will be packed individually and sent to pathologists who are blind to the method sequence.
  Arms: Group C
Procedure: Slow-pull, wet suction, standard suction — Patients will be sampled for a total of 3 consecutive FNA passes with a sequential method of "slow-pull", "wet suction", and "standard suction". After completing all the passes, the obtained specimen will be packed individually and sent to pathologists who are blind to the method sequence.
  Arms: Group D
Procedure: Wet suction, standard suction, slow-pull — Patients will be sampled for a total of 3 consecutive FNA passes with a sequential method of "wet suction", "standard suction", and "slow-pull". After completing all the passes, the obtained specimen will be packed individually and sent to pathologists who are blind to the method sequence.
  Arms: Group E
Procedure: Wet suction, slow-pull, standard suction — Patients will be sampled for a total of 3 consecutive FNA passes with a sequential method of "wet suction", "slow-pull", and "standard suction". After completing all the passes, the obtained specimen will be packed individually and sent to pathologists who are blind to the method sequence.
  Arms: Group F

SUMMARY:
The aim of this study is to compare endoscopic ultrasound guided-fine needle aspiration (EUS-FNA) with a standard 22-gauge needle using "standard suction", "slow-pull" and "wet suction" for thoracic/abdominal solid/solid-cystic lesions. Investigators intend to compare the effectiveness and safety of the three methods in order to discover the optimized technique for obtaining diagnostic material and making accurate diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* In-patients and out-patients between the age of 18years and 80 years with thoracic/abdominal solid/solid-cystic lesions for EUS-FNA.

Exclusion Criteria:

* Uncorrectable coagulopathy (INR > 1.5)
* Uncorrectable thrombocytopenia (platelet < 50,000)
* Cystic lesions
* Inaccessible lesions to EUS
* Contraindications for conscious sedation
* Uncooperative patients
* Refusal to consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of standard suction technique | 1 year
  A positive diagnosis of malignancy by an EUS biopsy specimen is accepted as a true positive. A benign diagnosis is confirmed by surgical tissue samples when available or clinical follow-up after 1 year.
Diagnostic yield of slow-pull technique | 1 year
  A positive diagnosis of malignancy by an EUS biopsy specimen is accepted as a true positive. A benign diagnosis is confirmed by surgical tissue samples when available or clinical follow-up after 1 year.
Diagnostic yield of wet suction technique | 1 year
  A positive diagnosis of malignancy by an EUS biopsy specimen is accepted as a true positive. A benign diagnosis is confirmed by surgical tissue samples when available or clinical follow-up after 1 year.
Specimen quality score of standard suction | Immediate
  EUS-FNA obtained specimen is scored as follows: 1) blood contamination: 0 for severe, 1 for moderate, 2 for few; 2) tissue structure: 0 for none, 1 for 1-2 structures seen, 2 for more than 3 structures seen; 3) cell quantity: 0 for <10/High power field(HPF), 1 for <50/HPF, 2 for >50/HPF; 4) diagnosability: 0 for hard to diagnose, 1 for suspicious diagnose, 2 for definite diagnosis.
Specimen quality score of slow-pull | Immediate
  EUS-FNA obtained specimen is scored as follows: 1) blood contamination: 0 for severe, 1 for moderate, 2 for few; 2) tissue structure: 0 for none, 1 for 1-2 structures seen, 2 for more than 3 structures seen; 3) cell quantity: 0 for <10/HPF, 1 for <50/HPF, 2 for >50/HPF; 4) diagnosability: 0 for hard to diagnose, 1 for suspicious diagnose, 2 for definite diagnosis.
Specimen quality score of wet suction | Immediate
  EUS-FNA obtained specimen is scored as follows: 1) blood contamination: 0 for severe, 1 for moderate, 2 for few; 2) tissue structure: 0 for none, 1 for 1-2 structures seen, 2 for more than 3 structures seen; 3) cell quantity: 0 for <10/HPF, 1 for <50/HPF, 2 for >50/HPF; 4) diagnosability: 0 for hard to diagnose, 1 for suspicious diagnose, 2 for definite diagnosis.

SECONDARY OUTCOMES:
Adverse event | 1 week
  Including bleeding, infection, pneumonia, perforation and other procedure related adverse events.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Qilu Hospital, Shandong University, Jinan, Shandong
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No